CLINICAL TRIAL: NCT00964041
Title: Effects of Weekly Dosing of D-cycloserine on Cognitive Function in Individuals With Schizophrenia.
Brief Title: Once Weekly D-cycloserine for Schizophrenia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Donald C. Goff, MD, Director of the Schizophrenia Clinical and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-P-001341; P50MH060450 (NIH); DATR A3-NSC
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Schizophrenia
Keywords: Cognitive Impairment; Neuroplasticity; D-cycloserine; N-methyl-D-aspartate (NMDA); Anti-Bacterial Agents; Mental Disorders; Psychotic Disorders; Antitubercular Agents; Schizophrenia and Disorders with Psychotic Features; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction; Mental Disorders; Psychotic Disorders; Schizophrenia Spectrum and Other Psychotic Disorders | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-cycloserine (Experimental): Participants will receive D-cycloserine weekly, one hour before any assessments, for eight weeks.
  Interventions: Drug: D-cycloserine
- Placebo (Placebo Comparator): Participants will receive placebo weekly, one hour before any assessments, for eight weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-cycloserine — 50 mg by mouth weekly, one hour before assessments, for eight weeks.
  Other Names: Seromycin; Cycloserine
  Arms: D-cycloserine
Drug: Placebo — Placebo by mouth, weekly, one hour before any assessments, each week for eight weeks.
  Arms: Placebo

SUMMARY:
This is a parallel-group, placebo-controlled trial examining the cognitive effects at weeks 1, 4, & 8 of once-weekly oral D-cycloserine 50 mg added to a stable dose of antipsychotic for 8 weeks in adult outpatients with schizophrenia.

DETAILED DESCRIPTION:
In a previous placebo-controlled trial, investigators demonstrated significant improvement of negative symptoms with once-weekly D-cycloserine treatment. In addition, investigators found significant improvement of memory consolidation following the first dose; however, the effect on memory consolidation was lost after several weeks. The "practice effect" of weekly measurement of memory consolidation using repeated administration of the Logical Memory Test may have resulted in a "ceiling effect" which would obscure drug/placebo differences. In the current study, investigators propose to administer the Logical Memory Test at four-week intervals (weeks 1, 4 and 8) to avoid the ceiling effect. Additionally a measurement will be added of negative symptoms at week 4 to better characterize the time course of negative symptom improvement.

Hypotheses:

1. Assess the effects of a single dose of D-cycloserine 50 mg on memory consolidation as measured by the Logical Memory Test compared to placebo.
2. Assess the persistence of once-weekly D-cycloserine effects on memory consolidation measured at weeks 4 & 8.
3. Assess the effects of repeated weekly dosing of D-cycloserine on performance on a standard cognitive battery at week 8 compared to placebo.
4. Assess effects of weekly D-cycloserine dosing on negative symptoms at weeks 4 & 8 compared to placebo.
5. Assess tolerability and side effects of weekly D-cycloserine compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age 18-65 years
3. Diagnosis of schizophrenia or schizoaffective disorder, depressed type
4. Stable dose of antipsychotic for at least 4 weeks.
5. Able to provide informed consent
6. Able to complete a cognitive battery

Exclusion Criteria:

1. Current treatment with clozapine
2. Dementia
3. Seizure disorder
4. Unstable medical illness
5. Active substance abuse
6. Pregnancy, nursing, or unwilling to use appropriate birth control measures during participation if female and fertile.
7. Severe renal insufficiency (Serum creatinine > 1.5 mg/dL)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Effect of repeated weekly dosing of D-cycloserine on performance on a standard cognitive battery. | Baseline (Week 0) and End of Study (Week 8)

SECONDARY OUTCOMES:
Effects of weekly D-cycloserine dosing on negative symptoms at weeks 4 & 8 compared to placebo. | Baseline (Week 0) and End of Study (Week 8)
Effect of a single dose of D-cycloserine 50 mg on memory consolidation as measured by the Logical Memory Test compared to placebo. | Same Day (Single Dose - Week 1)
Assess the persistence of once-weekly D-cycloserine effects on memory consolidation measured at weeks 4 & 8. | Week 4 and Week 8
Assess tolerability and side effects of weekly D-cycloserine compared to placebo | Weekly measurements for 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Donald C Goff, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States